# A Brief Virtual ACT Workshop for Emotional Eating Study Protocol Di Sante, Frayn & Knäuper

June 11th 2020

## Methodology/Procedures

- 1. **Recruitment:** Advertisements will be placed in McGill University's staff newsletter with an e-mail address for interested participants contact the research team via a given e-mail address. Explanations of the workshop and research study will be sent to interested participants and different timeslots will be offered. Interested participants will be asked to list their availabilities in order of preference so that they may be assigned into groups. They will be sent a confirmation e-mail with the date of the workshop and a link to an online questionnaire (baseline questionnaire) which will include the consent form.
- 2. **Baseline assessments:** All participants will read the consent form (and agree to participate using a checkbox), and complete a demographics questionnaire, the DEBQ-EE, the Distress Tolerance Scale (DTS; Simons & Gaher, 2005), the Food Acceptance and Awareness Questionnaire (FAAQ; Juarascio, Forman, Timko, Butryn, & Goodwin, 2011), and the Mindful Eating Questionnaire (MEQ; Framson et al., 2009) prior to attending the workshop. They will also be asked a series of questions pertaining to values clarification and commitment in relation to emotional eating. Finally, they will be asked to complete two additional items recording the number of times they engaged in emotional eating as well as how much often they were able to stop emotional eating after starting. These items were developed by the authors. All questionnaires will be completed online through Qualtrics.
- 3. **Intervention:** Workshops will be 3 hours in length (delivered over the course of 2, 1.5h sessions held 1-week apart) and held via the Zoom online platform on different dates. They will be facilitated by the author of the workshop manual, Mallory Frayn, a clinical psychology PhD candidate. The intervention will be modeled after Frayn et al.'s (2019) intervention, which was a 1-day ACT workshop derived from Forman et al.'s (2013) "Mind

Your Health program". During the workshop, the following topics will be discussed, based on the three processes of ACT relevant to emotional eating identified in Forman and Butryn's (2014) review:

#### Session 1

- (1) Values Clarification and Commitment
  - a. Exploring values and why it is important for participants to reduce their emotional eating.
    Values clarification will be emphasized to allow participants to identify that emotional eating is inconsistent with values pertaining to health and wellness. This values clarification will set the framework for motivating alternative, value- consistent behaviours.
  - b. Using values to make decisions and to engage in committed action (teaching the BOLD technique and walking participants through examples). Participants will be asked to brainstorm alternative, value-consistent behaviours that do not involve eating.

## (2) Acceptance/Distress Tolerance

a. Introducing acceptance, specifically acceptance of negative emotions, within the ACT model (e.g., use tug-of-war metaphor and dropping the rope to elucidate this). Using acceptance in the context of emotional eating to explain that participants do not have to respond to their negative emotions by eating.

## (3) Mindfulness/Awareness applied to emotions

a. Introducing mindfulness for emotional awareness. Using awareness of physical sensations related to emotions, with an emphasis on the separation of thoughts and physical sensations related to emotions, to help recognize emotional arousal in the context of emotional eating.

#### **Session 2**

## (1) Acceptance/Distress Tolerance

a. Introducing the concept of urge surfing, allowing participants to normalize cravings that arise as a result of negative emotions. Teaching participants concrete steps to employ urge surfing to sit with negative emotions and cravings, rather than acting on them by eating.

# (2) Mindfulness/Awareness applied to eating

- a. Introducing mindful eating and mindfulness of hunger/satiety signals. Participants will be asked to participate in an exercise where they are taught to mindfully eat a chosen food that they will have on hand. Mindful eating will be applied to emotional eating, as emotional eating is typically a mindless experience. Participants will be encouraged to pay mindful awareness of their hunger/satiety cues, and eat mindfully in a way that is physically and psychologically satisfying. An overview of hunger/satiety signal awareness and monitoring will be provided.
- (3) Program review, habit formation, and commitment to values
  - a. Following the introduction and application of these three techniques, a discussion will be held to review what was taught and to identify which techniques resonate most with participants. The facilitator will answer/clarify any questions people may have about any of the concepts taught. Towards the end of the second session, the facilitator will also introduce the concept of habit formation and the importance of practicing the techniques such that they become automatic. The workshop will conclude with committed action, bringing the discussion back to the commitment to values discussed at beginning of session.

4. **Post-intervention, 2-weeks and 3-month follow-ups:** At these time points, participants will be asked to complete the same battery of questionnaires they completed prior to taking the workshop. The purpose of these follow-up assessments is to assess changes in these variables from baseline to post-intervention, 2-weeks and 3-months post-intervention to examine the effectiveness of the workshop in the short and long term.

#### References

- Forman, E. M., & Butryn, M. L. (2014). A new look at the science of weight control: How acceptance and commitment strategies can address the challenge of self-regulation.

  Appetite, 84, 171-180.
- Forman, E. M., Butryn, M. L., Juarascio, A. S., Bradley, L. E., Lowe, M. R., Herbert, J. D., & Shaw, J. A. (2013). The mind your health project: A randomized controlled trial of an innovative behavioral treatment for obesity. *Obesity*, *21*, 1119-1126.
- Framson, C., Kristal, A. R., Schenk, J. M., Littman, A. J., Zeliadt, S., & Benitez, D. (2009).

  Development and validation of the mindful eating questionnaire. *Journal of the American Dietetic Association*, 109(8), 1439-1444.
- Frayn, M., Khanyari, S., & Knäuper, B. (2019). A 1-day acceptance and commitment therapy workshop leads to reductions in emotional eating in adults. *Eating and Weight Disorders-Studies on Anorexia*, *Bulimia and Obesity*, 1-13.
- Juarascio, A., Forman, E., Timko, A., Butryn, M., & Goodwin, C. (2011). The development and validation of the food craving acceptance and action questionnaire (FAAQ). *Eating Behaviors*, *12*, 182-187.
- Simons, J. S., & Gaher, R. M. (2005). The Distress Tolerance Scale: Development and validation of a self-report measure. *Motivation and Emotion*, *29*, 83-102.
- van Strien, T., Frijters, J., Bergers, G., & Defares, P. B. (1986). The Dutch Eating Behavior Questionaire (DEBQ) for assessment of restrained, emotional, and external eating behavior. *International Journal of Eating Disorders*, *5*, 295-315.